CLINICAL TRIAL: NCT04081623
Title: Trans-abdominal Fetal Pulse Oximetry: Signal Integrity
Status: Terminated | Type: Observational
Why Stopped: COVID-19
Sponsor: Raydiant Oximetry, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ROSS Gen 2
Record Dates: First submitted 2019-09-03; First posted 2019-09-09 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Fetal Distress
MeSH Terms: conditions — Fetal Distress

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Clinic: This group is undergoing their scheduled visit for Non-Stress Test (NST) or Biophysical Profile (BPP)
  Interventions: Device: Raydiant Oximetry Sensing System
- Labor and Delivery: This group is in active labor.
  Interventions: Device: Raydiant Oximetry Sensing System

INTERVENTIONS:
Device: Raydiant Oximetry Sensing System — The investigational device is used to record fetal pulse signals.
  Other Names: ROSS

SUMMARY:
This project is set up to advance and integrate the established mathematical principles of oxygen saturation to model with increasing accuracy the "body in a body" problem of fetus in mother; similar to existing pulse oximeters,

DETAILED DESCRIPTION:
The investigational device is a non-invasive fetal pulse oximeter that measures fetal arterial pulse signal using safe, noninvasive, transabdominal near-infrared spectroscopy. The optical sensor will obtain fetal pulse oximetry signals. Women will also undergo sonographic evaluation to assess distance from maternal skin to fetal tissue and to confirm fetal presentation and position. There is no change to standard of care procedures for fetal heart rate monitoring. The fetal heart rate that will be monitored with the investigational device will be used for research purposes only. Results will not be used to guide or alter patient management.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women with singleton pregnancies, vertex presentation
2. Age ≥ 18 years
3. Healthy women ≥ 28 weeks gestation undergoing either Non-Stress test (NST) or Biophysical profile (BPP) OR
4. Healthy women ≥ 37 weeks in labor
5. Vertex presentation

Exclusion Criteria:

1. Age <18 years
2. Multiple gestation ( twins, triplets)
3. Presentation other than vertex
4. < 28 weeks of gestation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: Women undergoing their scheduled visit to the MFM clinic for a NST/BPP or in latent labor
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2019-04-16 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
Fetal signal integrity | During NST, BPP, or active labor
  Integrity of the fetal signal relative to background maternal signal and biologic/electronic noise, and related to fetal position, presentation and the depth of the fetus from maternal skin.

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No